CLINICAL TRIAL: NCT03814512
Title: Improving Insulin Resistance and Energy Metabolism Through Sleep Extension in Adolescents: The REM Study
Brief Title: Improving Insulin Resistance and Energy Metabolism Through Sleep Extension in Adolescents
Acronym: REM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-2396
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sleep; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a pilot study testing the intervention arm of the RCT. No control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extended Sleep Intervention (ES) (Experimental): Participants will receive a Standard Care Diet and Physical Activity Education Intervention (SC) and an Extended Sleep Intervention (ES). For the SC, participants will have their diet, physical activity, and screen time assessed by study interventionist. Prescribed goals will be determined collaboratively through discussion with participants and parents. For the ES, participants will subsequently be prescribed a sleep schedule that allows them to obtain 1.5 h more time in bed compared to their typical sleep. Prescribed bedtimes and wake times will be determined collaboratively.
  Interventions: Behavioral: Extended Sleep Intervention

INTERVENTIONS:
Behavioral: Extended Sleep Intervention — Participants will receive an Extended Sleep Intervention (ES). Participants will be prescribed a sleep schedule that allows them to obtain approximately 1.5 h more time in bed compared to their typical sleep. Prescribed bedtimes and wake times will be determined collaboratively through discussion with participants and parents.

SUMMARY:
The investigators propose to deliver a 4-week sleep extension intervention to adolescents to evaluate feasibility of the protocol and obtain preliminary data on intra-individual changes in metabolic parameters induced by sleep extension.

DETAILED DESCRIPTION:
The specific aims of this feasibility study are to 1) examine the feasibility of recruitment and retention of adolescents with overweight/obesity, pre-diabetes, and inadequate sleep into a sleep extension intervention; 2) assess adherence of a sleep extension intervention to increase total sleep time in adolescents with overweight/obesity, pre-diabetes, and inadequate sleep; 3) determine estimates of mean and variability of potential intervention outcomes including metabolomic, body composition, and substrate oxidation. The investigators propose to deliver a 4-week sleep extension intervention to adolescents to evaluate feasibility of the protocol and obtain preliminary data on intra-individual changes in metabolic parameters induced by sleep extension.

This proposal is the first step to demonstrate feasibility in delivering the intervention in a research setting, measure the effect of the intervention on changing sleep duration, and examine changes in obesity-related IR metabolites that would lead to improved IR in an adolescent population with pre-diabetes. The long-term goal is to disseminate an effective and feasible T2D prevention program that can be sustainably implemented in clinical weight management settings.

ELIGIBILITY:
Inclusion Criteria:

1. High school students between the age of 13-19 years
2. BMI >85th percentile for age and sex
3. Prediabetes defined as a HbA1c 5.7-6.4%
4. Tanner Stage 4-5 (based on breast development for girls and testicular size for boys)

Exclusion Criteria:

1. Any medications that affect insulin resistance or sleep (e.g., metformin, stimulants, atypical antipsychotics, current use of oral steroids)
2. Regular use of melatonin or other sleep aids
3. A prior diagnosis of a sleep disorder (e.g. insomnia, delayed sleep phase syndrome, obstructive sleep apnea) or abnormal scores on sleep disorders screening measures
4. Type 2 diabetes (HbA1c ≥ 6.5%)
5. IQ<70 or severe mental illness that may impact sleep or ability to consent/assent (e.g., schizophrenia, psychotic episodes), verified through chart review
6. Teens not enrolled in a traditional high school academic program (e.g., home school students)
7. Schedules that would preclude participants from adhering to the sleep extension protocol (e.g. night shift employment)
8. Travel across more than two time zones in the 2 weeks prior to the study

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Total Sleep Time | up to 12 weeks
  The amount of time (hours:minutes) the participant sleeps post-intervention compared to pre-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Lafayette, Colorado, United States

IPD SHARING:
Plan to Share IPD: No